CLINICAL TRIAL: NCT00397644
Title: Enhancing a Medical Home for Vulnerable Children by Addressing Family Psychosocial Problems at Well-Child Care Visits: THE WE CARE Project
Brief Title: Assisting Low-Income Families at Pediatric Well-Child Care Visits
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Collaborators: The Commonwealth Fund (Other)
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 20060351
Record Dates: First submitted 2006-11-07; First posted 2006-11-09 (Estimated); Last update posted 2023-11-01 (Actual); Status verified 2023-10

CONDITIONS: Low-income Children's Well-child Care Visit
Keywords: pediatrician; well-child care visit; low-income children; family psychosocial problem
MeSH Terms: interventions — Surveys and Questionnaires

INTERVENTIONS:
Behavioral: Prompting (survey instrument/resources list) (behavior)

SUMMARY:
The objective of this study is to evaluate the impact and feasibility of a practice-based intervention on the discussion and referral of family psychosocial topics at well-child care visits at a medical home for low-income children.

DETAILED DESCRIPTION:
Many low-income families have family psychosocial problems such as unemployment, housing difficulties, and food insecurity. Pediatric guidelines that pediatricians should be discussing and assisting these families. However, to date few routine do. The primary hypotheses for this study is that the WE CARE (Well-child care visit, Evaluation, Community resources, Advocacy, Referral, Education)intervention would increase the discussion and referral rates for family psychosocial problems at well-child care visits.

ELIGIBILITY:
Inclusion Criteria:

* Caregivers of children aged 2 months to 10 years who present for well-child care visit at a pediatric clinic

Exclusion Criteria:

* Non-English speaking
* Foster parents
* Previously enrolled parent
* No access to telephone

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 200
Dates: Start 2006-03; Study Completion 2006-06

PRIMARY OUTCOMES:
Discussion of family psychosocial problem
Referral of family psychosocial problem
Contacting community resources

CONTACTS AND LOCATIONS:
Overall Officials: Arvin Garg, MD, MPH, Principal Investigator — Johns Hopkins School of Medicine; Janet Serwint, MD, Principal Investigator — Johns Hopkins School of Medicine
Locations (1):
- Harriet Lane Clinic at Johns Hopkins Hospital, Baltimore, Maryland, United States

REFERENCES:
- [Derived] Kalra N, Hooker L, Reisenhofer S, Di Tanna GL, Garcia-Moreno C. Training healthcare providers to respond to intimate partner violence against women. Cochrane Database Syst Rev. 2021 May 31;5(5):CD012423. doi: 10.1002/14651858.CD012423.pub2. PMID 34057734
- [Derived] Garg A, Butz AM, Dworkin PH, Lewis RA, Thompson RE, Serwint JR. Improving the management of family psychosocial problems at low-income children's well-child care visits: the WE CARE Project. Pediatrics. 2007 Sep;120(3):547-58. doi: 10.1542/peds.2007-0398. PMID 17766528